CLINICAL TRIAL: NCT02414763
Title: Pilot Study of a Brief Intervention for Medically Hospitalized Suicide Attempt Survivors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Western Kentucky University (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 131757
Record Dates: First submitted 2014-12-16; First posted 2015-04-13 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Suicide Attempt
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care as Usual (No Intervention): Participants will receive usual care services provided to suicide attempt survivors, including inpatient psychiatry, outpatient psychotherapy, and case management.
- Teachable Moment Brief Intervention (Experimental): The brief intervention consists of engaging the patient in conversation regarding suicidal ambivalence (desire to live vs. desire to die), collaborative discovery of primary and secondary drivers of suicidality, functional analysis of the suicidal ideation and behaviors, and crisis response planning. Participants will also receive usual care services provided to suicide attempt survivors, including inpatient psychiatry, outpatient psychotherapy, and case management.
  Interventions: Behavioral: Teachable Moment Brief Intervention

INTERVENTIONS:
Behavioral: Teachable Moment Brief Intervention — functional analysis, collaborative interpersonal style
  Arms: Teachable Moment Brief Intervention

SUMMARY:
The current study proposes to study the feasibility and acceptability of a brief psychosocial intervention delivered to suicide attempt survivors hospitalized on a medical/surgical floor or inpatient psychiatry unit at Vanderbilt University Medical Center. The proposed study will involve training of care providers affiliated with Vanderbilt University Medical Center to deliver the brief intervention. Additionally, the participants will complete baseline, 1, 3, and 12-month assessments on outcomes of interest, including readiness to change problematic behaviors, engagement in outpatient mental health services, suicidal ideation, self-harming behavior, and reasons for living.

DETAILED DESCRIPTION:
One-hundred participants will be recruited from a medical/surgical floor or inpatient psychiatry unit at Vanderbilt University Medical Center. The PI, other Attending Psychiatrists, Psychiatry Resident Physicians, Clinical Psychology Trainees, Psychiatric Nurse Practitioners, Psychiatric Social Workers, and Psychiatric Nurse Case Managers will serve as study therapists. A member from the Vanderbilt University research team will obtain informed consent for the participants and then administer the baseline assessment battery. Patients will then be randomized to either (1) a group receiving care as usual plus an experimental intervention targeting suicidal thoughts and behaviors or to (2) a group receiving care as usual. Patients randomized to the experimental group will receive the intervention prior to discharge from the medical center, most likely on the same day as the baseline assessment battery. Patients receiving the experimental intervention will then be asked to complete a brief post-intervention client satisfaction survey. All study participants will then complete telephone follow-up assessments at 1, 3, and 12 months. The intervention will consist of no more than 90 minutes of 1:1 interaction with a study clinician. The baseline assessment battery will take approximately 30 minutes, the post-intervention measures will take approximately 10 minutes, and the 1-, 3-, and 12-month assessment batteries will take approximately 30 minutes. Maximum length of time in the study is approximately 3.75 hours.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above
* Inpatient on medical/surgical unit either currently or prior to transfer to inpatient psychiatric unit
* Admitted following a suicide attempt
* Sufficient English to benefit from psychotherapy in English
* Consents to be a research participant

Exclusion Criteria:

* Lack of sufficient English to participate in psychotherapy in English
* Prisoner/inmate at time of admission
* Too cognitively impaired, delirious, or psychotic to respond to psychotherapeutic intervention before end of stay in the medical center. Determination of cognitive impairment, delirium, agitation, and psychosis will be determined through the referral phone call between discussions with research team members and the Adult Psychiatry Consultation Service Physician providing care to the patient, as well as the interventionist's own clinical assessment of the patient at the outset of the brief intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-07; Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | Immediately following Brief Intervention
  The 8-item Client Satisfaction Questionnaire is a general measure of individual satisfaction with health and human services that takes 3-8 minutes to complete.

SECONDARY OUTCOMES:
Change in Stages of Change Questionnaire | Baseline, 1-, 3-, and 12-months interviews
  The Stages of Change Questionnaire is an 18-item measure based on the original, 32- item scale created by McConnaughy, Prochaska, and Verlicer. The measure has shown acceptable levels of internal consistency in an adult sample (α = .75 to .87) and predictive validity of response to treatment.
Change in Scale for Suicide Ideation | Baseline, 1-, 3-, and 12-months interviews
  The Scale for Suicide Ideation is a 19-item assessment used to evaluate the current intensity of the patient's specific attitudes toward, behavior, and plans to commit suicide. The measure has been the primary outcome measure in several trials targeting suicidal patients and has evidence of strong psychometrics
Change in Suicide Attempt Self-Injury Count | Baseline, 1-, 3-, and 12-months interviews
  The Suicide Attempt Self-Injury Count is a brief two-page instrument determining for the first, most recent, and most severe suicide attempt or non-suicidal self-injury (SASI) the date, method of SASI attempt used in index and previous attempts according to the definitions of Linehan et al. (e.g., using definitions of self-inflicted injuries which include situations of actual tissue damage and situations where tissue damage would have occurred except for outside intervention or sheer luck [e.g., firearm jammed]), intent to die (i.e., intent to die, ambivalent, no intent to die), highest level of medical treatment received, and lethality.
Change in Interpersonal Needs Questionnaire | Baseline, 1-, 3-, and 12-months interviews
  The Interpersonal Needs Questionnaire is a 25-item measure that inquires about the extent to which individuals feel connected to others (i.e., belongingness) and the extent to which they feel like a burden on the people in their lives (i.e., perceived burdensomeness). The measure has been used in previous research examining mechanisms underlying suicide attempt survivors and has demonstrated acceptable psychometric properties
Change in Reasons for Living Inventory | Baseline, 1-, 3-, and 12-months interviews
  The Reasons for Living Inventory is a 48-item measure that rates the importance of different reasons why people choose not to kill themselves. It has shown strong internal consistency and test-retest reliability
Change in Health Services and Medication Use | 1-, 3-, and 12-months interviews
  The Health Services and Medication Use measure will be utilized to examine history of mental health services and medication use in lifetime, previous year, and previous month time periods. The measure was developed and utilized in the National Study of Costs and Outcomes for Trauma.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen S O'Connor, Ph.D., Principal Investigator — Western Kentucky University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] O'Connor SS, Mcclay MM, Choudhry S, Shields AD, Carlson R, Alonso Y, Lavin K, Venanzi L, Comtois KA, Wilson JE, Nicolson SE. Pilot randomized clinical trial of the Teachable Moment Brief Intervention for hospitalized suicide attempt survivors. Gen Hosp Psychiatry. 2020 Mar-Apr;63:111-118. doi: 10.1016/j.genhosppsych.2018.08.001. Epub 2018 Aug 10. PMID 30389316